CLINICAL TRIAL: NCT05683184
Title: Characterization of CB1 Receptors Using [11-C]OMAR in Opioid Use Disorder
Brief Title: OMAR Opioid Use Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Anahita Bassir Nia, Assistant Professor of Psychiatry, Yale University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000033525; 1R21DA052864-01A1 (NIH); 2K12DA000167-31 (NIH)
Record Dates: First submitted 2022-12-20; First posted 2023-01-13 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Healthy Control; Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — 4-cyano-1-(2,4-dichlorophenyl)-5-(4-methoxyphenyl)-N-(piperidin-1-yl)-1H-pyrazole-3-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Other): Healthy volunteers with no current or past major medical or psychiatric history
  Interventions: Drug: [11C]OMAR
- Opioid Use Disorder (Other): Patients diagnosed with opioid use disorder
  Interventions: Drug: [11C]OMAR

INTERVENTIONS:
Drug: [11C]OMAR — For each [11C]OMAR PET scan, up to 20 mCi of [11C]OMAR will be administered.
  Other Names: [11C] JHU75528

SUMMARY:
The goal of this research study is to examine the endocannabinoid (eCB) function in vivo in individuals with opioid use disorder (OUD) by measuring cannabinoid receptor 1 (CB1R) availability.

DETAILED DESCRIPTION:
The investigators will image brain cannabinoid receptors using Positron Emission Tomography (PET) imaging and the radioligand [11C] OMAR, in healthy individuals and individuals diagnosed with opioid use disorder. Research participants may complete screening, MRI, PET scan and follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Male and female 18 years and older
* DSM-5 diagnosis of opioid use disorder (for OUD group)
* Physically healthy i.e., no clinically unstable medical conditions
* Written informed consent and have capacity to consent and comply with study procedures

Exclusion Criteria:

* Current neuro-psychiatric illness or severe systemic disease (opioid use disorder is permitted in the OUD group).
* Presence of ferromagnetic metal in the body or heart pacemaker
* Have had exposure to ionizing radiation that in combination with the study tracer would result in a cumulative exposure that exceeds recommended exposure limits
* Are claustrophobic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
CB1R Availability | One time within 4 weeks of screening
  To compare cortical CB1R availability in individuals diagnosed with opioid use disorder on chronic methadone maintenance vs. matched healthy controls.

SECONDARY OUTCOMES:
Serum Endocannabinoid Levels | One time within 4 weeks of screening
  To explore group differences in serum endocannabinoid levels in individuals diagnosed with opioid use disorder on chronic methadone maintenance vs. matched healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Anahita Bassir Nia, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, Clinical Neuroscience Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No